CLINICAL TRIAL: NCT03551678
Title: Novel Strategies to Combat Post-Traumatic Osteoarthritis (PTOA): Gait Retraining to Reduce Joint Loading, Inflammation, and PTOA Risk
Brief Title: Gait Retraining to Reduce Joint Loading, Inflammation, and PTOA Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Constance Chu, MD, Study Principal Investigator, VA Palo Alto Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46025; CDMRP-PR171647 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Gait retraining (Experimental): Eight weeks of active-feedback gait retraining. The gait retraining device measures pressure/force under the lateral side of the foot and activates vibration if loading crosses a set threshold. The location of the vibration is customized for each subject to achieve maximal sensitivity.
  Interventions: Device: Active feedback gait retraining

INTERVENTIONS:
Device: Active feedback gait retraining — The device measures pressure/force under the lateral side of the foot and activates vibration if loading crosses a set threshold. The location of the vibration is customized for each subject to achieve maximal sensitivity.

SUMMARY:
The purpose of this study is to determine changes to knee joint loading, biological markers, and cartilage structure following a novel active feedback gait retraining program in anterior cruciate ligament reconstructed patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years
* history of primary ACLR with or without meniscal repair
* full weight-bearing status
* neutral to varus knee alignment
* plans to remain in the area for at least 8 months.

Exclusion Criteria:

* Kellgren-Lawrence (KL) radiographic grade > 2
* additional injury or surgery to the involved knee
* BMI >30 kg/m2
* use of walking, orthopedic, or prosthetic assistive device
* pregnancy
* inability to have MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Adduction Moment | Change from baseline to immediately after 8 weeks of retraining
  Knee Joint Loading (%Bw*Ht) will be assessed at baseline and immediately after gait retraining

SECONDARY OUTCOMES:
Medial knee compartment qMRI | Change from baseline to 6 months after retraining
  Changes to quantitative MRI measures at 6 months after retraining will be correlated with changes to joint loading
Knee Adduction Moment | Change from baseline to 3 months after retraining
  Knee Joint Loading (%Bw*Ht)
Knee Adduction Moment | Change from baseline to 6 months after retraining
  Knee Joint Loading (%Bw*Ht)
Serum inflammatory markers | Change from baseline to immediately after 8 weeks of retraining
  Changes to serum inflammatory markers immediately after the end of training from baseline will be correlated with changes to joint loading

CONTACTS AND LOCATIONS:
Overall Officials: Constance Chu, MD, Principal Investigator — VAPAHCS and Stanford University
Locations (1):
- VA Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No